CLINICAL TRIAL: NCT03230864
Title: Interventional, Randomized, Double-blind, Active-controlled Study of the Efficacy of Lu AF35700 in Patients With Early-in-disease or Late-in-disease Treatment-resistant Schizophrenia
Brief Title: Efficacy of Lu AF35700 in Patients With Early-in-disease or Late-in-disease Treatment-resistant Schizophrenia
Acronym: Anew
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: New data; the study was terminated based on new efficacy data from another study
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17303A
Record Dates: First submitted 2017-07-24; First posted 2017-07-27 (Actual); Results first posted 2020-01-07 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Treatment-resistant Schizophrenia
Keywords: Treatment-resistant schizophrenia; Lu AF35700
MeSH Terms: conditions — Schizophrenia, Treatment-Resistant | interventions — Lu AF35700; Risperidone; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Prospective Confirmation (PC) Period (Experimental): Single (patient)-blinded treatment period with risperidone or olanzapine for 6 weeks
  Interventions: Drug: Risperidone; Drug: Olanzapine
- Double-blind treatment (DBT) period, Lu AF35700 10 mg (Experimental): Eligible patients from PC period (based on criteria to which investigator and patient are blinded ), will be randomly assigned (1:1) double-blind treatment in DBT period, 8 weeks
  Interventions: Drug: Lu AF35700
- DBT Period, Continued treatment from PC Period (Experimental): Eligible patients from PC period (based on criteria to which investigator and patient are blinded ), will be randomly assigned (1:1) double-blind treatment in DBT period, 8 weeks. Patients in this arm will continue with the same treatment and dose as at the last visit of the PC Period
  Interventions: Drug: Risperidone; Drug: Olanzapine

INTERVENTIONS:
Drug: Lu AF35700 — 10 mg/day, encapsulated tablets, orally
  Arms: Double-blind treatment (DBT) period, Lu AF35700 10 mg
Drug: Risperidone — 4-6 mg/day, encapsulated tablets, orally
  Arms: DBT Period, Continued treatment from PC Period; Prospective Confirmation (PC) Period
Drug: Olanzapine — 15-20 mg/day, encapsulated tablets, orally
  Arms: DBT Period, Continued treatment from PC Period; Prospective Confirmation (PC) Period

SUMMARY:
This study evaluates the efficacy of 10 mg/day Lu AF35700 on symptoms of schizophrenia in patients with early-in-disease (ED) or late-in-disease (LD) treatment-resistant schizophrenia (TRS)

DETAILED DESCRIPTION:
In the study, patients will receive risperidone (4-6 mg/day), or, if recently failed on risperidone, olanzapine (15-20mg/day). Later during the study, patients will be randomized to either receive Lu AF35700 (10 mg/day), or continue their treatment from the prospective confirmation (PC) period.

The study consists of a Screening Period (up to 3 weeks), a single-blind PC Period (6 weeks), a Double-blind Treatment (DBT) Period (8 weeks), and a Safety Follow-up Period (6 weeks).

Patients who did not fulfil the randomization criteria for the DBT Period, were withdrawn from the study after the PC period.

Patients who fulfilled the randomization criteria for the DBT Period, continued into the DBT period and were randomized into one of the 2 treatmetn arms (1:1) with either Lu AF35700 10 mg or to continue the treatment allocated in the PC period (olanzapine or risperidone) at the dose set at the last visit of the PC period. This means that approximately half of the confirmed treatment-resistant patients were randomised back to the failed treatment in the PC period.

Data was not collected seperately for the DBT olanzapine and DBT risperidone participants, and there was no intent to compare Lu AF35700 to each drug seperately.

ELIGIBILITY:
Inclusion Criteria:

* The patient has schizophrenia, diagnosed according to DSM-5(TM). (Diagnostic and Statistical Manual of Mental Disorders) and confirmed by the Mini International Neuropsychiatric Interview for Schizophrenia and Psychotic Disorders (MINI-Schz).
* The patient is receiving treatment with a psychiatrist in either an inpatient or outpatient facility.
* The patient has been treated with adequate dose(s) of antipsychotic drug treatment for at least 2 weeks prior to the Screening Visit.
* The patient has failed to show an adequate response in the level of psychotic symptoms during at least one documented treatment trial with an adequate dose of an antipsychotic drug prescribed for an adequate time (at least lasting for 6 weeks) within 2 years prior to the Screening Visit. The failure to respond to the current antipsychotic drug treatment trial may be considered a retrospective failed treatment, if the patient has been treated for 6 weeks with adequate dose(s) of antipsychotic drug(s).
* The patient has a PANSS total score of ≥80 (on 1-7 scale) and a score of ≥4 (≥ "Moderate" on 1-7 scale) on at least 2 of the following PANSS items at the Screening and at Baseline 1 [Week 0] Visits: P2 - Conceptual disorganization, P3 - Hallucinatory behavior, P6 - Suspiciousness/persecution, G9 - Unusual thought content; AND the patient has a CGI-S score of ≥4 (≥ "Moderately ill") at the Screening and at Baseline 1 (Week 0) Visits.

Exclusion Criteria:

* The patient has any current primary psychiatric disorder other than schizophrenia, as assessed using the MINI-Schz.
* The patient suffers from mental retardation, organic mental disorders, or mental disorders due to a general medical condition (DSM-5™ criteria).
* The patient is experiencing an acute exacerbation of his/her psychotic symptoms.
* The patient has been treated with, AND is resistant to, clozapine according to the investigator's judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2018-12-23 (Actual); Study Completion 2019-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H.Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (41):
- United States (10):
  - University of California San Diego Health System, San Diego, California
  - Emory University Cognitive Neurology Clinic & ADRC, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Corrigan Mental Health Center, Fall River, Massachusetts
  - University Of Massachusetts Medical Center, Worcester, Massachusetts
  - Michigan Clinical Research Institute PC, Ann Arbor, Michigan
  - Kalamazoo Community Mental Health and Substance Abuse Services, Kalamazoo, Michigan
  - PsychCare Consultants Research, St Louis, Missouri
  - Creighton University, Omaha, Nebraska
  - Psychiatric and Behavioral Solutions, Salt Lake City, Utah
- Bulgaria (7):
  - SPH - Kardzhali, Kardzhali
  - State Psychiatric Hospital, Novi Iskar
  - UMHAT, Pleven
  - State Psychiatric Hospital, Radnevo
  - DCC St. Vrach and St.St. Kuzma and Damian, Sofia
  - MHC - Sofia, Sofia
  - MHAT - Targovishte, Targovishte
- Japan (10):
  - Takeda General Hospital - JP0009, Aizu-Wakamatsu
  - Takeda General Hospital, Fukushima
  - Kohnodai Hospital, Ichikawa
  - Nara Medical University Hospital, Kashihara
  - Sankeikai Nishigahara Hospital - JP0008, Kita-ku
  - University of Occupational and Environmental Health Hospital, Kitakyushu
  - National Center of Neurology and Psychiatry, Kodaira
  - Satokai Yuge Hospital, Kumamoto
  - NHO Ryukyu Hospital, Kunigami
  - Fujita Health University Hospital, Toyoake
- Russia (9):
  - GUZ Lipetsk Regional psychoneurological Hospital 1, Lipetsk
  - Lipetsk Regional Psychoneurological Hospital, Lipetsk
  - City Psychiatric Hospital # 6, Saint Petersburg
  - Psychoneurological Dispensary #10, Saint Petersburg
  - Psychoneurological Dispensary #1, Saint Petersburg
  - Samara Psychiatric Hospital, Samara
  - Tomsk National Research Medical Centre of the Russian Academy of Sciences, Tomsk
  - Yaroslavl Regional Clinical Psychiatric Hospital, Yaroslavl
  - Sverdlovsk Regional Clinical Psychiatric Hospital, Yekaterinburg
- United Kingdom (5):
  - Royal Edinburgh Hospital, Edinburgh
  - The Maudsley Hospital - GB0001, London
  - The Maudsley Hospital, London
  - Manchester Mental Health & Social Care NHS Trust - GB0003, Manchester
  - Manchester Mental Health & Social Care NHS Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients who did not fulfil the randomization criteria for the DBT period, were withdrawn from the study after the PC period. Patients who fulfilled the randomization crietria for the DBT period, continued into the DBT period. Patients randomized into the DBT period with risperidone or olanzapine were analyzed as one arm.
Groups:
- Prospective Confirmation (PC) Period, Risperidone: Single (patient)-blinded treatment period with risperidone or olanzapine for 6 weeks
  Risperidone: 4-6 mg/day, encapsulated tablets, orally
- PC Period, Olanzapine: Single (patient)-blinded treatment period with risperidone or olanzapine for 6 weeks
  Olanzapine: 15-20 mg/day, encapsulated tablets, orally
- Double-blind (DBT), Lu AF35700 10 mg: Lu AF35700: 10 mg/day, encapsulated tablets, orally for 8 weeks
- DBT, Continued Treatment From PC Period: Patients in this arm will continue the treatment allocated in the PC period at the dose set at the last visit of the PC period. The analysis is made independent on which treatment the patient was done (risperidone or olanzapine). 8 weeks treatment.
Period: Prospective Confirmation (PC) Period
Arm/Group | Prospective Confirmation (PC) Period, Risperidone | PC Period, Olanzapine | Double-blind (DBT), Lu AF35700 10 mg | DBT, Continued Treatment From PC Period
Started | 68 | 51 | 0 | 0
Completed | 36 | 32 | 0 | 0
Not Completed | 32 | 19 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 1 | 0 | 0
Not completed — Did not fulfill rand criteria DBT | 14 | 5 | 0 | 0
Not completed — Sponsor Decision | 9 | 9 | 0 | 0
Not completed — Study Personnel Decision | 1 | 0 | 0 | 0
Period: Double Blind Treatment (DBT) Period
Arm/Group | Prospective Confirmation (PC) Period, Risperidone | PC Period, Olanzapine | Double-blind (DBT), Lu AF35700 10 mg | DBT, Continued Treatment From PC Period
Started | 0 | 0 | 35 | 33
Completed | 0 | 0 | 27 | 31
Not Completed | 0 | 0 | 8 | 2
Not completed — Adverse Event | 0 | 0 | 5 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1
Not completed — Sponsor Decision | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Non-randomized Patients: Patients not randomized to double-blind treatment period, i.e. withdrawn from the study during or after the PC period, were analyzed as one arm, independent of treatment
- Double-blind Treatment (DBT) Period, Lu AF35700 10 mg: Lu AF35700: 10 mg/day, encapsulated tablets, orally for 8 weeks
- DBT, Continued Treatment From PC Period: Patients in this arm continued with the same treatment and dose as at the last visit of the PC period. Patients randomized into the DBT period with risperidone or olanzapine were analyzed as one arm independent of treatment.
- Total: Total of all reporting groups
Arm/Group | Non-randomized Patients | Double-blind Treatment (DBT) Period, Lu AF35700 10 mg | DBT, Continued Treatment From PC Period | Total
Number analyzed (Participants) | 51 | 35 | 33 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (12.53) | 42.9 (11.26) | 42 (12.26) | 42.5 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 15 | 17 | 55
  Male | 28 | 20 | 16 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 2 | 6
  Not Hispanic or Latino | 50 | 32 | 30 | 112
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 3 | 3 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 0 | 2 | 10
  White | 38 | 31 | 27 | 96
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2
PANSS total score [Mean (Standard Deviation); unit: units on a scale] — Positive and Negative Syndrome Scale (PANNS) total score administered by the investigator. It included a total of 30 items that evaluated the Positive Symptoms subscale, the Negative Symptoms subscale, the General Psychopathology subscale. Each item is rated from 1 (symprom not present) to 7 (symptom extremely severe). PANNS total score was calculated as sum of all items on the scale and ranged from 30 to 210. A higher score corresponded to a worse severity of schizophrenia.
  units on a scale | 98.1 (10.78) | 102.3 (12) | 101.6 (11.95) | 100.3 (11.54)
CGI-S score [Mean (Standard Deviation); unit: units on a scale] — CGI-S provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (Normal - not at all ill) to 7 (among the most extremely ill patients).
  units on a scale | 4.8 (0.64) | 4.8 (0.57) | 4.9 (0.55) | 4.82 (0.59)

OUTCOME MEASURES:

1. Primary Outcome: Change From Randomization to Week 8 in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: PANSS total score administered by the investigator. It included a total of 30 items that evaluated the Positive Symptoms subscale, the Negative Symptoms subscale, the General Psychopathology subscale. Each item is rated from 1 (symptom not present) to 7 (symptom extremely severe). PANSS total score was calculated as sum of all the items on the scale and ranged from 30 to 210. A negative score indicates an improvement compared to Randomization.
Time Frame: From Randomization to Week 8
Population: Only patients randomized to receive double-blind treatment in the DBT period are analyzed. Patients randomized into the DBT period with risperidone or olanzapine were analyzed as one arm. Overall Number of Participants Analysed is number of patients in the full-analysis set (FAS) with a week 8 observation
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- DBT, Continued Treatment From PC Period: Patients in this arm will continue on the same treatment and dose as at the last visit of the PC period (olanzapine or risperidone)
Arm/Group | Double-blind Treatment (DBT) Period, Lu AF35700 10 mg | DBT, Continued Treatment From PC Period
Number analyzed (Participants) | 27 | 31
units on a scale | -4.71 (2.22) | -10.19 (2.16)
Statistical Analysis 1: Comparison: Double-blind Treatment (DBT) Period, Lu AF35700 10 mg vs DBT, Continued Treatment From PC Period; The mean changes from randomization in PANNS total score was analysed using a mixed model for repeated measures (MMRM) approach. The model will include the fixed, categorical effects of treatment, strata, visit, treatment-by-visit interaction, fixed covariates of baseline scores and baseline scores-by-visit interaction. An unstructured (co)variance structure will be used to model the within-patient errors. The Kenward-Roger approximation will be used to estimate denominator degrees of freedom; Test type: Superiority; p = 0.0809, Mixed Model Repeated Measures; Mean Difference (Final Values) = 5.47, 95% CI 2-sided [-0.70 to 11.65]

2. Secondary Outcome: Change From Randomization to Week 8 in Global Clinical Impression - Severity of Illness (CGI-S) Score
Description: CGI-S provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (normal - not at all ill) to 7 (among the most extremely ill patients). Higher scores indicate worsening
Time Frame: From Randomization to Week 8
Population: Only patients randomized to receive double-blind treatment in the DBT period are analyzed. Patients randomized into the DBT period with risperidone or olanzapine were analyzed as one arm. Overall Number of Participants Analysed is number of patients in the FAS with a week 8 observation
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- DBT, Lu AF35700 10 mg: 10 mg encapsulated tablets administered orally, once daily.
  Lu AF35700: 10 mg/day, encapsulated tablets, orally
- DBT, Continued Treatment: Patients in this arm will continue on the same treatment and dose as at the last visit of the PC period (olanzapine or risperidone)
Arm/Group | DBT, Lu AF35700 10 mg | DBT, Continued Treatment
Number analyzed (Participants) | 27 | 31
units on a scale | -0.18 (0.12) | -0.37 (0.11)

3. Secondary Outcome: Change From Randomization to Week 8 in 16-item Negative Symptom Assessment (NSA-16 Total) Score
Description: The NSA-16 is a clinician-rated scale designed to assess the presence, severity, and range of negative symptoms associated with schizophrenia. The NSA-16 consists of 16 items arranged in 5 subdomains: communication dysfunction (items 1 to 4), emotional/affective dysfunction (items 5 to 7), dysfunction in sociality (items 8 to 10), motivational/hedonic dysfunction (items 11 to 14), and reduced psychomotor activity (items 15 and 16), and a Global Negative Symptom Rating. NSA-16 items are rated on a 6-point scale from 1 (behaviour is normal) to 6 (behaviour severely reduced), and a score of 9 if the item is not-rateable. The Global Negative Symptom Rating is rated from 1 (no evidence of symptoms) to 7 (extremely severe symptoms). The 16 items are summed to yield a total score ranging from 16 to 96 and the global rating ranges from 1 to 7.
Time Frame: From Randomization to Week 8
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | DBT, Lu AF35700 10 mg | DBT, Continued Treatment
Number analyzed (Participants) | 27 | 31
units on a scale | -2.99 (1.64) | -3.14 (1.58)

4. Secondary Outcome: Change From Randomization to Week 8 in PANSS Marder Negative Factor Score
Description: The PANSS Negative Factor score is a subset of the PANSS assessing negative symptoms of schizophrenia. The factor consist of the seven items: blunted affect, emotional withdrawal, poor rapport, passive social withdrawal, lack of spontaneity, motor retardation, and active social avoidance which are each rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS Negative Factor score (7 items) range from 7 to 49 with a higher score indicating greater severity of symptoms.
Time Frame: From Randomization to Week 8
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | DBT, Lu AF35700 10 mg | DBT, Continued Treatment
Number analyzed (Participants) | 27 | 31
units on a scale | -1.51 (0.77) | -1.74 (0.75)

5. Secondary Outcome: Response
Description: Response is defined as a ≥20% reduction in PANSS total score from Randomization
Time Frame: at Week 8
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | DBT, Lu AF35700 10 mg | DBT, Continued Treatment
Number analyzed (Participants) | 27 | 31
Participants | 6 | 13

ADVERSE EVENTS:
Time Frame: 20 weeks
Groups:
- Prospective Confirmation (PC) Period - Risperidone; PC Period - Olanzapine: Patients not randomized to double-blind treatment
- Double Blind Treatment (DBT) Period - Lu AF35700 10 mg: Lu AF35700: 10 mg/day, encapsulated tablets, orally for 8 weeks
- DBT Period, Continued Treatment From PC Period: Patients in this arm continued with the same treatment and dose as at the last visit of the PC Period. This arm is analyzed as one single treatment arm independent on which treatment was administered (olanzapine or risperidone for 8 weeks).
Arm/Group | Prospective Confirmation (PC) Period - Risperidone | PC Period - Olanzapine | Double Blind Treatment (DBT) Period - Lu AF35700 10 mg | DBT Period, Continued Treatment From PC Period
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/51 | 0/35 | 0/33
Serious Adverse Events (participants affected / at risk) | 1/68 | 1/51 | 0/35 | 0/33
Other Adverse Events (participants affected / at risk) | 16/68 | 3/51 | 8/35 | 7/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prospective Confirmation (PC) Period - Risperidone (N=68) | PC Period - Olanzapine (N=51) | Double Blind Treatment (DBT) Period - Lu AF35700 10 mg (N=35) | DBT Period, Continued Treatment From PC Period (N=33)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prospective Confirmation (PC) Period - Risperidone (N=68) | PC Period - Olanzapine (N=51) | Double Blind Treatment (DBT) Period - Lu AF35700 10 mg (N=35) | DBT Period, Continued Treatment From PC Period (N=33)
Weight increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Akathisia (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 6 (7) | 1 (1) | 4 (4) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4) | 0 (0) | 1 (1) | 2 (2)
Schizophrenia (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early and hence the statistical analysis was conducted on a smaller sample size than originally planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-09-07): https://cdn.clinicaltrials.gov/large-docs/64/NCT03230864/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/64/NCT03230864/SAP_001.pdf